CLINICAL TRIAL: NCT05070793
Title: Improving Alcohol Use Disorder Treatment for Gender Minority Populations
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional Research Pause
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeremy D. Kidd, MD, MPH, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7953; 1K23AA028296 (NIH)
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
Keywords: transgender; gender minority; gender identity; interpersonal; psychotherapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Culturally adapted interpersonal psychotherapy (Other): Individual psychotherapy intervention based on Brief Interpersonal Psychotherapy (IPT-B) with additional cultural adaptation for transgender and nonbinary individuals.
  Interventions: Behavioral: Culturally adapted interpersonal psychotherapy

INTERVENTIONS:
Behavioral: Culturally adapted interpersonal psychotherapy — Individual psychotherapy based on Brief Interpersonal Psychotherapy, culturally adapted for transgender and nonbinary individuals.

SUMMARY:
Gender minority (GM; transgender and gender non-conforming) individuals experience disproportionately high rates of hazardous drinking and alcohol use disorder (AUD) and are an NIH-designated disparity population (NOT-MD-19-001). Despite marked disparities and unique alcohol risk factors, there are no evidence-based alcohol interventions for this population. This study will conduct mixed-methods formative research with an established multi-site longitudinal GM cohort to develop and assess the feasibility of the first culturally-adapted psychosocial treatment intervention for GMs with AUD. The study will evaluate an adapted version of interpersonal psychotherapy (IPT), with adaptations intended to enhance the responsiveness of IPT to the unique life experiences of GM individuals that may influence alcohol consumption.

DETAILED DESCRIPTION:
BACKGROUND

Transgender and nonbinary individuals (TGNB; i.e., gender minorities) have a gender identity and/or gender expression that differs from the female or male sex that they were assigned at birth. This difference (gender incongruence) can cause psychological distress. Comprising roughly 0.5% of the U.S. population, TGNB people bear numerous health disparities including hazardous drinking (HD; binge drinking and/or heavy drinking) and alcohol use disorder (AUD). These relate to stigma and discrimination. Numerous studies have found high rates of past 30-day drinking (21-58%), binge drinking (21-51%), and heavy drinking (26%). These rates exceed general population estimates of past 30-day binge drinking (16.3%) and heavy drinking (5.9%).

TGNB people suffer interpersonal disruptions that serve as culturally-distinct alcohol risk factors. Such interpersonal disruptions are related to HD via increased interpersonal distress. TGNB people have interpersonal distress in unique contexts such as gender transition and anti-TGNB discrimination/stigma. Gender transition is the process of reducing gender incongruence through aesthetics (e.g., clothing), hormones (e.g., estrogen/testosterone), and/or surgery (e.g., vaginoplasty/phalloplasty). This often brings changes in key interpersonal relationships, varying from renegotiation (e.g., a heterosexual couple adjusting to being a same-gender couple after one partner transitions) to dissolution (e.g., divorce). TGNB people also experience high rates of discrimination (distal minority stress) that affect relationships (e.g., a biased employer). In both contexts, interpersonal disruptions and distress increase alcohol risk, possibly via diminished social support. Many TGNB adults report drinking to cope with interpersonal stressors. Conversely, TGNB peer support protects against such distress and HD.

Culturally-adapted treatment may benefit interpersonal disruptions and distress occurring in the context of discrimination. Of TGNB adults, 24% reported having to teach their healthcare providers about TGNB experiences. Studies of addiction treatment staff found that most knew little about TGNB issues and nearly half held negative or ambivalent views about TGNB patients. Qualitative studies of TGNB individuals in addiction treatment found stigmatization was common, including prohibitions on disclosing TGNB identity or being forced to wear clothing inconsistent with gender identity. This can lead to treatment avoidance or termination.

Cultural-adaptation considers "language, culture, and context" to increase treatment compatibility with patients' cultural norms/values. Among various cultural adaptation models, the Cultural Sensitivity Framework (CSF) was specifically designed for addiction research. In CSF, adaptation addresses both surface (concrete) and deep (abstract) structures. In racial/ethnic and sexual minority (lesbian/gay/bisexual) studies, cultural adaptation improved treatment acceptability, retention, and effectiveness; including for addiction. Aside from conceptual discussions, there are no culturally-adapted TGNB AUD interventions.

Separate evidence-based approaches exist for interpersonal distress (e.g., IPT) and alcohol (e.g., motivation interviewing; MI), but there are no integrated treatments for both that target the interpersonal contexts TGNB people face. IPT, a time-limited manualized psychotherapy, identifies an interpersonal problem area (grief, role disputes, role transitions, interpersonal deficits) and reduces symptoms by enhancing interpersonal coping and social support. IPT's focus on "role transition" and "role disputes" especially applies to gender transition-related interpersonal disruptions and distress. Over 133 clinical trials have validated IPT for depression and for PTSD-common co-morbidities for TGNB individuals. IPT AUD research is limited. Extant research on co-morbid depression and AUD is equivocal, but these studies were designed with depression as the primary outcome and enrolled mostly non-TGNB patients with low-level drinking. Researchers have called for studies of IPT with MI strategies for AUD in populations with salient interpersonal risk factors (i.e., TGNB populations).

STUDY PROCEDURES

Overall strategy: This pilot trial of culturally-adapted Brief Interpersonal Psychotherapy (IPT-B) for transgender and nonbinary (TGNB) individuals with AUD utilizes a single-arm, pre-post, convergent mixed methods design to explore whether and how the intervention engages interpersonal targets. This design enables the investigators to link qualitative themes regarding individuals' experiences of the intervention with quantitative measures of interpersonal targets. The investigators will also evaluate the feasibility of research and intervention procedures and the acceptability of the information and support provided by the therapist.

Participants: TGNB individuals with alcohol use disorder (AUD) (N = 20). We anticipate enrolling 50% individuals assigned female at birth and at least 30% non-White individuals.

Screening: Interested individuals will be complete a standardized telephone interview and will be invited to participate if they meet eligibility criteria for an evaluation. This subsequent evaluation will include the MINI International Neuropsychiatric Interview(57) to assess current and lifetime DSM-5 diagnoses, a psychiatric and medical evaluation (including urine drug screen). Eligible individuals will be invited to enroll in the trial and will provide written informed consent. Individuals will be compensated for this screening evaluation.

Assessment Schedule: After baseline assessment, there will be 9 weekly intervention visits plus 1-month follow-up. The intervention will be delivered by trained clinical staff. At intervention completion, participants will be provided with referrals for continued outpatient treatment and a list of Alcoholics Anonymous meetings. Study staff will administer outcomes measures without participating in intervention delivery. This will include administering alcohol and interpersonal target measures at Baseline, Weeks 5 and 9, and 1-month follow-up. At intervention completion (Week 9), study staff will administer acceptability measures; including qualitative assessment of treatment acceptability, interpersonal targets, and drinking. Participants will be compensated for completing study assessments. Psychotherapy will not be compensated. For safety, study staff will obtain vital signs and a breathalyzer before each visit; and will assess alcohol withdrawal and overall symptom severity at each visit. Staff will also assess for suicide risk and psychiatric symptoms at Baseline, Weeks 5 and 9, and 1-month follow-up.

Measures:

Feasibility: Staff will track data pertaining to recruitment, retention, and assessment procedures following CONSORT guidelines; including the duration and number of intervention contacts per participant.

Acceptability: After each session, therapists and participants will complete the Working Alliance Inventory-Short Form (WAI-SF) to assess their perception of the therapeutic alliance. Staff will use the Treatment Acceptability Questionnaire (TAQ) to assess participants' perceptions of the intervention's clarity/helpfulness/appropriateness/relevance and the therapist's skill and trustworthiness. This will include open-ended, qualitative questions about participants' experiences of the intervention (e.g., culturally-tailored elements); including perceived strengths and weaknesses, session length/content, therapeutic alliance, value of TGNB cultural adaptations, and recommendations for improvement.

Fidelity: Staff will audio record all intervention sessions. Sessions will be randomly chosen and reviewed by the Principal Investigator and an IPT research expert. Sessions will be scored using the Collaborative Study Psychotherapy Rating Scale-Form 6.

Demographics: Staff will collect information about age, race/ethnicity, assigned sex, education, and annual household income. Staff will also assess current/lifetime gender-affirming hormone use and surgeries.

Discrimination and Stigma: For descriptive purposes, staff will assess experiences of discrimination with the Everyday Discrimination Scale and stigma with the Stigma Consciousness Questionnaire.

Alcohol Consumption: The Timeline Followback (TLFB; 28-day at baseline; 7-day thereafter) to assess drinking and urine ethyl glucuronide (EtG), a metabolite of alcohol metabolism, as a biomarker of recent (~past 24-hour) drinking.

Alcohol Motivation/Expectancy: Readiness to Change Questionnaire-Treatment Version (RCQ-TV) to measure motivation to reduce drinking, Coping Strategies Scale (CSS) for coping ability with alcohol cravings, Alcohol Abstinence Self-Efficacy Scale (AASE) to measure participants' perceived ability to reduce drinking, Alcohol Expectancy Questionnaire (AEQ) to assess anticipated positive alcohol experiences, and Drinker Inventory of Consequences (DrInC) to measure negative alcohol consequences.

Interpersonal Targets: The Multidimensional Scale of Perceived Social Support (MSPSS) for family/friend support, an adapted scale from AFFIRM for GM peer support, the Social Adjustment Scale-Self Report (SAS-SR) to assess satisfaction with social supports, and the Inventory of Interpersonal Problems (IIP) to assess interpersonal disruptions/distress. Staff will use the Reflective Functioning Questionnaire (RFQ) to measure mentalization (ability to understand mental states of oneself and others). Increased mentalization capacity may be one mechanism by which IPT reduces interpersonal distress and psychiatric symptoms.

Co-morbidities: The Hamilton Depression Rating Scale (HAM-D) and PTSD Checklist (PCL-5) will assess these symptom domains. I will assess concurrent drug use with the Timeline Followback (28-day at baseline; 7-day thereafter) and urine qualitative drug screens.

Safety: Breathalyzer to assess alcohol intoxication, the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) to evaluate alcohol withdrawal, the Columbia Suicide Severity Rating Scale (CSSRS) for suicide risk, and the Clinical Global Impressions Scale for severity (CGI-S) and improvement (CGI-I).

Data analysis: This trial's purpose is to collect preliminary data about feasibility and engagement of interpersonal targets.

Missed Visits/Drop-Out: These rates are reported directly as part of the primary feasibility outcome.

Hypotheses: At least 75% of participants will complete the intervention (feasibility); At least 80% will report treatment satisfaction (acceptability).

Primary Analysis: Primary outcomes will be treatment feasibility (% completion) and acceptability (Treatment Acceptability Questionnaire). We will report quantitative data using descriptive statistics. For qualitative data, interviews will be audio recorded and professionally transcribed. Next, transcripts will be iteratively coded, identifying codes and categories (codebook) that we will apply to the entire data set. To ensure consistency, we will double-code 10% of interviews.

Exploratory outcomes: While this study does not have statistical power to test formal hypotheses regarding alcohol outcomes or interpersonal targets, we will examine % reduction in heavy drinking days (≥5 drinks for GM women; ≥4 for GM men) and % days abstinent as well as alcohol motivation/expectancy and interpersonal target variables. WE will measure pre-post change and report these using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* GM self-identification
* English fluency,
* Current DSM-5 Alcohol use disorder (AUD) (moderate-to-severe)
* AUD treatment-seeking
* Able to give informed consent and comply with study procedures

Exclusion Criteria:

* Severe psychiatric symptoms that would interfere with treatment (e.g., psychosis, active suicidality)
* History of severe alcohol withdrawal (e.g., seizure, delirium tremens)
* Legally mandated to treatment
* Current DSM-5 SUD other than alcohol/nicotine/caffeine/cannabis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Completing all study sessions | 9 weeks
  Percentage of participants who complete all intervention sessions
Acceptability - Treatment Acceptability Questionnaire | 9 weeks
  Treatment Acceptability Questionnaire

SECONDARY OUTCOMES:
Heavy drinking days | 9 weeks and 13 weeks
  Percent reduction in heavy drinking days (≥5 drinks for GM women; ≥4 for GM men)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Kidd, MD, Principal Investigator — New York State Psychiatric Institute/Research Foundation for Mental Hygiene, Inc
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all IPD that underlie results in publications related the primary and secondary hypotheses of the trial.
Time Frame: Starting 6 months after publication
Access Criteria: All requests will be reviewed by the Principal Investigator. Expectation will be that requests have accompanying IRB approval for analysis of de-identified data.

REFERENCES:
- [Background] Bockting W. From construction to context: Gender through the eyes of the transgendered. SIECUS Report. 1999;28(1):3-5.
- [Background] Institute of Medicine (US) Committee on Lesbian, Gay, Bisexual, and Transgender Health Issues and Research Gaps and Opportunities. The Health of Lesbian, Gay, Bisexual, and Transgender People: Building a Foundation for Better Understanding. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK64806/ PMID 22013611
- [Background] Meyer IH, Brown TN, Herman JL, Reisner SL, Bockting WO. Demographic Characteristics and Health Status of Transgender Adults in Select US Regions: Behavioral Risk Factor Surveillance System, 2014. Am J Public Health. 2017 Apr;107(4):582-589. doi: 10.2105/AJPH.2016.303648. Epub 2017 Feb 16. PMID 28207334
- [Background] Blosnich JR, Marsiglio MC, Dichter ME, Gao S, Gordon AJ, Shipherd JC, Kauth MR, Brown GR, Fine MJ. Impact of Social Determinants of Health on Medical Conditions Among Transgender Veterans. Am J Prev Med. 2017 Apr;52(4):491-498. doi: 10.1016/j.amepre.2016.12.019. Epub 2017 Feb 1. PMID 28161034
- [Background] U.S. Department of Health and Human Services. Healthy People 2020: Lesbian, Gay, Bisexual, and Transgender Health. 2014 [Available from: https://www.healthypeople.gov/2020/topics-objectives/topic/lesbian-gay-bisexual-and-transgender-health.
- [Background] James SE, Herman JL, Rankin S, Kiesling M, Mottet L, Anafi M. The Report of the 2015 U.S. Transgender Survey Washington, D.C.: National Center for Transgender Equality; 2016 [Available from: https://transequality.org/sites/default/files/docs/usts/USTS-Full-Report-Dec17.pdf.
- [Background] Bockting WO, Miner MH, Swinburne Romine RE, Hamilton A, Coleman E. Stigma, mental health, and resilience in an online sample of the US transgender population. Am J Public Health. 2013 May;103(5):943-51. doi: 10.2105/AJPH.2013.301241. Epub 2013 Mar 14. PMID 23488522
- [Background] Coulter RW, Blosnich JR, Bukowski LA, Herrick AL, Siconolfi DE, Stall RD. Differences in alcohol use and alcohol-related problems between transgender- and nontransgender-identified young adults. Drug Alcohol Depend. 2015 Sep 1;154:251-9. doi: 10.1016/j.drugalcdep.2015.07.006. Epub 2015 Jul 16. PMID 26210734
- [Background] Santos GM, Rapues J, Wilson EC, Macias O, Packer T, Colfax G, Raymond HF. Alcohol and substance use among transgender women in San Francisco: prevalence and association with human immunodeficiency virus infection. Drug Alcohol Rev. 2014 May;33(3):287-95. doi: 10.1111/dar.12116. Epub 2014 Mar 14. PMID 24628655
- [Background] Gilbert PA, Pass LE, Keuroghlian AS, Greenfield TK, Reisner SL. Alcohol research with transgender populations: A systematic review and recommendations to strengthen future studies. Drug Alcohol Depend. 2018 May 1;186:138-146. doi: 10.1016/j.drugalcdep.2018.01.016. Epub 2018 Mar 10. PMID 29571076
- [Background] Martinez O, Wu E, Levine EC, Munoz-Laboy M, Spadafino J, Dodge B, Rhodes SD, Rios JL, Ovejero H, Moya EM, Baray SC, Carballo-Dieguez A, Fernandez MI. Syndemic factors associated with drinking patterns among Latino men and Latina transgender women who have sex with men in New York City. Addict Res Theory. 2016;24(6):466-476. doi: 10.3109/16066359.2016.1167191. Epub 2016 Apr 10. PMID 28077938
- [Background] Rowe C, Santos GM, McFarland W, Wilson EC. Prevalence and correlates of substance use among trans female youth ages 16-24 years in the San Francisco Bay Area. Drug Alcohol Depend. 2015 Feb 1;147:160-6. doi: 10.1016/j.drugalcdep.2014.11.023. Epub 2014 Dec 15. PMID 25548025
- [Background] Scheim AI, Bauer GR, Shokoohi M. Heavy episodic drinking among transgender persons: Disparities and predictors. Drug Alcohol Depend. 2016 Oct 1;167:156-62. doi: 10.1016/j.drugalcdep.2016.08.011. Epub 2016 Aug 11. PMID 27542688
- [Background] Centers for Disease Control and Prevention. BRFSS Prevalence and Trends Data 2015 [Available from: https://www.cdc.gov/brfss/brfssprevalence/index.html.
- [Background] Kidd JD, Jackman KB, Wolff M, Veldhuis CB, Hughes TL. Risk and Protective Factors for Substance Use among Sexual and Gender Minority Youth: A Scoping Review. Curr Addict Rep. 2018 Jun;5(2):158-173. doi: 10.1007/s40429-018-0196-9. Epub 2018 May 26. PMID 30393591
- [Background] Bockting WO, Coleman E. Developmental stages of the transgender coming-out process: Toward an integrated identity. In: Ettner R, Monstrey S, Coleman E, editors. Principles of Transgender Medicine and Surgery. 2nd ed. New York, NY: Routledge; 2016. p. 137-258.
- [Background] Gonzalez CA, Gallego JD, Bockting WO. Demographic Characteristics, Components of Sexuality and Gender, and Minority Stress and Their Associations to Excessive Alcohol, Cannabis, and Illicit (Noncannabis) Drug Use Among a Large Sample of Transgender People in the United States. J Prim Prev. 2017 Aug;38(4):419-445. doi: 10.1007/s10935-017-0469-4. PMID 28405831
- [Background] World Professional Association for Transgender Health. Standards of Care for the Health of Transsexual, Transgender, and Gender Nonconforming People. 7th ed2011.
- [Background] Chester K, Lyons A, Hopner V. 'Part of me already knew': the experiences of partners of people going through a gender transition process. Cult Health Sex. 2017 Dec;19(12):1404-1417. doi: 10.1080/13691058.2017.1317109. Epub 2017 May 2. PMID 28463049
- [Background] Platt LF. An Exploratory Study of Predictors of Relationship Commitment for Cisgender Female Partners of Transgender Individuals. Fam Process. 2020 Mar;59(1):173-190. doi: 10.1111/famp.12400. Epub 2018 Oct 11. PMID 30311216
- [Background] Veldorale-Griffin A, Darling CA. Adaptation to Parental Gender Transition: Stress and Resilience Among Transgender Parents. Arch Sex Behav. 2016 Apr;45(3):607-17. doi: 10.1007/s10508-015-0657-3. Epub 2016 Jan 12. PMID 26758455
- [Background] Bockting W, Coleman E, Deutsch MB, Guillamon A, Meyer I, Meyer W 3rd, Reisner S, Sevelius J, Ettner R. Adult development and quality of life of transgender and gender nonconforming people. Curr Opin Endocrinol Diabetes Obes. 2016 Apr;23(2):188-97. doi: 10.1097/MED.0000000000000232. PMID 26835800
- [Background] Katz-Wise SL, Budge SL. Cognitive and interpersonal identity processes related to mid-life gender transitioning in transgender women. Couns Psychol Quart. 2015;28(2):150-74.
- [Background] Meyer IH. Prejudice, social stress, and mental health in lesbian, gay, and bisexual populations: conceptual issues and research evidence. Psychol Bull. 2003 Sep;129(5):674-697. doi: 10.1037/0033-2909.129.5.674. PMID 12956539
- [Background] Keuroghlian AS, Reisner SL, White JM, Weiss RD. Substance use and treatment of substance use disorders in a community sample of transgender adults. Drug Alcohol Depend. 2015 Jul 1;152:139-46. doi: 10.1016/j.drugalcdep.2015.04.008. Epub 2015 Apr 22. PMID 25953644
- [Background] Coulter RW, Birkett M, Corliss HL, Hatzenbuehler ML, Mustanski B, Stall RD. Associations between LGBTQ-affirmative school climate and adolescent drinking behaviors. Drug Alcohol Depend. 2016 Apr 1;161:340-7. doi: 10.1016/j.drugalcdep.2016.02.022. Epub 2016 Feb 23. PMID 26946989
- [Background] Pinto RM, Melendez RM, Spector AY. Male-to-Female Transgender Individuals Building Social Support and Capital From Within a Gender-Focused Network. J Gay Lesbian Soc Serv. 2008 Sep 1;20(3):203-220. doi: 10.1080/10538720802235179. PMID 20418965
- [Background] Staples JM, Neilson EC, George WH, Flaherty BP, Davis KC. A descriptive analysis of alcohol behaviors across gender subgroups within a sample of transgender adults. Addict Behav. 2018 Jan;76:355-362. doi: 10.1016/j.addbeh.2017.08.017. Epub 2017 Aug 18. PMID 28903090
- [Background] Pflum SR, Testa RJ, Balsam KF, Goldblum PB, Bongar B. Social support, trans community connectedness, and mental health symptoms among transgender and gender nonconforming adults. Psychol Sex Orientat Gend Divers. 2015;2(3):281-6.
- [Background] Valentine SE, Shipherd JC. A systematic review of social stress and mental health among transgender and gender non-conforming people in the United States. Clin Psychol Rev. 2018 Dec;66:24-38. doi: 10.1016/j.cpr.2018.03.003. Epub 2018 Mar 28. PMID 29627104
- [Background] Eliason MJ, Hughes T. Treatment counselor's attitudes about lesbian, gay, bisexual, and transgendered clients: urban vs. rural settings. Subst Use Misuse. 2004 Mar;39(4):625-44. doi: 10.1081/ja-120030063. PMID 15115216
- [Background] Mullens AB, Fischer J, Stewart M, Kenny K, Garvey S, Debattista J. Comparison of Government and Non-Government Alcohol and Other Drug (AOD) Treatment Service Delivery for the Lesbian, Gay, Bisexual, and Transgender (LGBT) Community. Subst Use Misuse. 2017 Jul 3;52(8):1027-1038. doi: 10.1080/10826084.2016.1271430. Epub 2017 Mar 20. PMID 28318357
- [Background] Lombardi E. Substance use treatment experiences of transgender/transsexual men and women. J LGBT Health Res. 2007;3(2):37-47. doi: 10.1300/J463v03n02_05. PMID 19835040
- [Background] Lyons T, Shannon K, Pierre L, Small W, Krusi A, Kerr T. A qualitative study of transgender individuals' experiences in residential addiction treatment settings: stigma and inclusivity. Subst Abuse Treat Prev Policy. 2015 May 7;10:17. doi: 10.1186/s13011-015-0015-4. PMID 25948286
- [Background] Bernal G, Jimenez-Chafey MI, Domenech Rodriguez MM. Cultural adaptation of treatments: A resource for considering culture in evidence-based practice. Prof Psychol-Res Pr. 2009;40:361-8. 36. Resnicow K, Soler R, Braithwaite RL, Ahluwalia JS, Butler J. Cultural sensitivity in substance use prevention. J Community Psychol. 2000;28(3):271-90.
- [Background] Barrera M Jr, Castro FG, Strycker LA, Toobert DJ. Cultural adaptations of behavioral health interventions: a progress report. J Consult Clin Psychol. 2013 Apr;81(2):196-205. doi: 10.1037/a0027085. Epub 2012 Jan 30. PMID 22289132
- [Background] Pearson CR, Kaysen D, Huh D, Bedard-Gilligan M. Randomized Control Trial of Culturally Adapted Cognitive Processing Therapy for PTSD Substance Misuse and HIV Sexual Risk Behavior for Native American Women. AIDS Behav. 2019 Mar;23(3):695-706. doi: 10.1007/s10461-018-02382-8. PMID 30607757
- [Background] Hernandez Robles E, Maynard BR, Salas-Wright CP, Todic J. Culturally adapted substance use interventions for Latino adolescents. Res Social Work Prac. 2018;28(7):789-801.
- [Background] Steinka-Fry KT, Tanner-Smith EE, Dakof GA, Henderson C. Culturally sensitive substance use treatment for racial/ethnic minority youth: A meta-analytic review. J Subst Abuse Treat. 2017 Apr;75:22-37. doi: 10.1016/j.jsat.2017.01.006. Epub 2017 Jan 23. PMID 28237051
- [Background] Valdez LA, Flores M, Ruiz J, Oren E, Carvajal S, Garcia DO. Gender and Cultural Adaptations for Diversity: A Systematic Review of Alcohol and Substance Abuse Interventions for Latino Males. Subst Use Misuse. 2018 Aug 24;53(10):1608-1623. doi: 10.1080/10826084.2017.1417999. Epub 2018 Jan 24. PMID 29364763
- [Background] Benish SG, Quintana S, Wampold BE. Culturally adapted psychotherapy and the legitimacy of myth: a direct-comparison meta-analysis. J Couns Psychol. 2011 Jul;58(3):279-89. doi: 10.1037/a0023626. PMID 21604860
- [Background] Baskerville NB, Dash D, Shuh A, Wong K, Abramowicz A, Yessis J, Kennedy RD. Tobacco use cessation interventions for lesbian, gay, bisexual, transgender and queer youth and young adults: A scoping review. Prev Med Rep. 2017 Feb 16;6:53-62. doi: 10.1016/j.pmedr.2017.02.004. eCollection 2017 Jun. PMID 28271021
- [Background] Pachankis JE, Hatzenbuehler ML, Rendina HJ, Safren SA, Parsons JT. LGB-affirmative cognitive-behavioral therapy for young adult gay and bisexual men: A randomized controlled trial of a transdiagnostic minority stress approach. J Consult Clin Psychol. 2015 Oct;83(5):875-89. doi: 10.1037/ccp0000037. Epub 2015 Jul 6. PMID 26147563
- [Background] Austin A, Craig SL, Alessi EJ. Affirmative Cognitive Behavior Therapy with Transgender and Gender Nonconforming Adults. Psychiatr Clin North Am. 2017 Mar;40(1):141-156. doi: 10.1016/j.psc.2016.10.003. Epub 2016 Dec 12. PMID 28159140
- [Background] Budge SL. Interpersonal psychotherapy with transgender clients. Psychotherapy (Chic). 2013 Sep;50(3):356-359. doi: 10.1037/a0032194. PMID 24000851
- [Background] Weissman MM, Markowitz JC, Klerman GL. The Guide to Interpersonal Psychotherapy. Oxford, UK: Oxford University Press; 2017.
- [Background] Johnson JE, Stout RL, Miller TR, Zlotnick C, Cerbo LA, Andrade JT, Nargiso J, Bonner J, Wiltsey-Stirman S. Randomized cost-effectiveness trial of group interpersonal psychotherapy (IPT) for prisoners with major depression. J Consult Clin Psychol. 2019 Apr;87(4):392-406. doi: 10.1037/ccp0000379. Epub 2019 Feb 4. PMID 30714749
- [Background] Weissman MM. Recent non-medication trials of interpersonal psychotherapy for depression. Int J Neuropsychopharmacol. 2007 Feb;10(1):117-22. doi: 10.1017/S1461145706006936. Epub 2006 Jun 20. PMID 16787556
- [Background] Krupnick JL, Melnikoff E, Reinhard M. A Pilot Study of Interpersonal Psychotherapy for PTSD in Women Veterans. Psychiatry. 2016 Spring;79(1):56-69. doi: 10.1080/00332747.2015.1129873. PMID 27187513
- [Background] Krupnick JL, Green BL, Stockton P, Miranda J, Krause E, Mete M. Group interpersonal psychotherapy for low-income women with posttraumatic stress disorder. Psychother Res. 2008 Sep;18(5):497-507. doi: 10.1080/10503300802183678. PMID 18816001
- [Background] Markowitz JC, Petkova E, Neria Y, Van Meter PE, Zhao Y, Hembree E, Lovell K, Biyanova T, Marshall RD. Is Exposure Necessary? A Randomized Clinical Trial of Interpersonal Psychotherapy for PTSD. Am J Psychiatry. 2015 May;172(5):430-40. doi: 10.1176/appi.ajp.2014.14070908. Epub 2015 Feb 13. PMID 25677355
- [Background] Nuttbrock L, Bockting W, Rosenblum A, Hwahng S, Mason M, Macri M, Becker J. Gender abuse, depressive symptoms, and substance use among transgender women: a 3-year prospective study. Am J Public Health. 2014 Nov;104(11):2199-206. doi: 10.2105/AJPH.2014.302106. Epub 2014 Sep 11. PMID 25211716
- [Background] Markowitz JC, Kocsis JH, Christos P, Bleiberg K, Carlin A. Pilot study of interpersonal psychotherapy versus supportive psychotherapy for dysthymic patients with secondary alcohol abuse or dependence. J Nerv Ment Dis. 2008 Jun;196(6):468-74. doi: 10.1097/NMD.0b013e31817738f1. PMID 18552624
- [Background] Gamble SA, Talbot NL, Cashman-Brown SM, He H, Poleshuck EL, Connors GJ, Conner KR. A pilot study of interpersonal psychotherapy for alcohol-dependent women with co-occurring major depression. Subst Abus. 2013;34(3):233-41. doi: 10.1080/08897077.2012.746950. PMID 23844953
- [Background] Brache K. Advancing interpersonal therapy for substance use disorders. Am J Drug Alcohol Abuse. 2012 Jul;38(4):293-8. doi: 10.3109/00952990.2011.643995. Epub 2012 Jan 13. PMID 22243427
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Janavs J, Weiller E, Keskiner A, et al. The validity of the Mini International Neuropsychiatric Interview (MINI) according to the SCID-P and its reliability. Eur Psychiat. 1997;12(5):232-41.
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Hatcher RL, Gillasby JA. Development and validation of a revised short version of the Working Alliance Inventory. Psychother Res. 2006;16(1):12-25.
- [Background] Hunsley J. Development of the Treatment Acceptability Questionnaire. J Psychopathol Behav. 1992;14(1):55-64.
- [Background] Amole MC, Cyranowski JM, Conklin LR, Markowitz JC, Martin SE, Swartz HA. Therapist Use of Specific and Nonspecific Strategies Across Two Affect-Focused Psychotherapies for Depression: Role of Adherence Monitoring. J Psychother Integr. 2017 Sep;27(3):381-394. doi: 10.1037/int0000039. Epub 2016 Jun 6. PMID 29225450
- [Background] Hill CE, O'Grady KE, Elkin I. Applying the Collaborative Study Psychotherapy Rating Scale to rate therapist adherence in cognitive-behavior therapy, interpersonal therapy, and clinical management. J Consult Clin Psychol. 1992 Feb;60(1):73-9. doi: 10.1037//0022-006x.60.1.73. PMID 1556289
- [Background] Williams DR, Yan Yu, Jackson JS, Anderson NB. Racial Differences in Physical and Mental Health: Socio-economic Status, Stress and Discrimination. J Health Psychol. 1997 Jul;2(3):335-51. doi: 10.1177/135910539700200305. PMID 22013026
- [Background] Pinel EC. Stigma consciousness: the psychological legacy of social stereotypes. J Pers Soc Psychol. 1999 Jan;76(1):114-28. doi: 10.1037//0022-3514.76.1.114. PMID 9972557
- [Background] Sobell LC, Sobell MB. Timeline Follow-Back: A technique for assessing self-reported alcohol consumption. In: Litten RZ, Allen JP, editors. Measuring Alcohol Consumption. Clifton, NJ: Humana; 1992. p. 41-72.
- [Background] Rollnick S, Heather N, Gold R, Hall W. Development of a short 'readiness to change' questionnaire for use in brief, opportunistic interventions among excessive drinkers. Br J Addict. 1992 May;87(5):743-54. doi: 10.1111/j.1360-0443.1992.tb02720.x. PMID 1591525
- [Background] Litt MD, Kadden RM, Cooney NL, Kabela E. Coping skills and treatment outcomes in cognitive-behavioral and interactional group therapy for alcoholism. J Consult Clin Psychol. 2003 Feb;71(1):118-28. doi: 10.1037//0022-006x.71.1.118. PMID 12602432
- [Background] DiClemente CC, Carbonari JP, Montgomery RP, Hughes SO. The Alcohol Abstinence Self-Efficacy scale. J Stud Alcohol. 1994 Mar;55(2):141-8. doi: 10.15288/jsa.1994.55.141. PMID 8189734
- [Background] Brown SA, Christiansen BA, Goldman MS. The Alcohol Expectancy Questionnaire: an instrument for the assessment of adolescent and adult alcohol expectancies. J Stud Alcohol. 1987 Sep;48(5):483-91. doi: 10.15288/jsa.1987.48.483. PMID 3669677
- [Background] Forcehimes AA, Tonigan JS, Miller WR, Kenna GA, Baer JS. Psychometrics of the Drinker Inventory of Consequences (DrInC). Addict Behav. 2007 Aug;32(8):1699-704. doi: 10.1016/j.addbeh.2006.11.009. Epub 2006 Dec 19. PMID 17182194
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Frost DM, Meyer IH. Measuring community connectedness among diverse sexual minority populations. J Sex Res. 2012;49(1):36-49. doi: 10.1080/00224499.2011.565427. Epub 2011 May 24. PMID 21512945
- [Background] Weissman MM, Olfson M, Gameroff MJ, Feder A, Fuentes M. A comparison of three scales for assessing social functioning in primary care. Am J Psychiatry. 2001 Mar;158(3):460-6. doi: 10.1176/appi.ajp.158.3.460. PMID 11229989
- [Background] Gude T, Moum T, Kaldestad E, Friis S. Inventory of interpersonal problems: a three-dimensional balanced and scalable 48-item version. J Pers Assess. 2000 Apr;74(2):296-310. doi: 10.1207/S15327752JPA7402_9. PMID 10879357
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Markowitz JC, Skodol AE, Bleiberg K. Interpersonal psychotherapy for borderline personality disorder: possible mechanisms of change. J Clin Psychol. 2006 Apr;62(4):431-44. doi: 10.1002/jclp.20242. PMID 16470711
- [Background] Hayden MC, Mullauer PK, Gaugeler R, Senft B, Andreas S. Improvements in mentalization predict improvements in interpersonal distress in patients with mental disorders. J Clin Psychol. 2018 Dec;74(12):2276-2286. doi: 10.1002/jclp.22673. Epub 2018 Jul 11. PMID 29998458
- [Background] Robinson SM, Sobell LC, Sobell MB, Leo GI. Reliability of the Timeline Followback for cocaine, cannabis, and cigarette use. Psychol Addict Behav. 2014 Mar;28(1):154-62. doi: 10.1037/a0030992. Epub 2012 Dec 31. PMID 23276315